CLINICAL TRIAL: NCT04981717
Title: A Randomized, Double-Blind, Placebo-Controlled Study in Cat-Allergic Patients With Allergic Rhinitis Who Live With a Cat to Assess the Efficacy and Safety of Anti-Fel d 1 Antibodies During Natural Cat Exposure in the Home
Brief Title: A Study to Examine the Efficacy and Safety of Anti-Fel d 1 Antibodies Injections in Cat-allergic Adolescent and Adult Patients With Allergic Rhinitis Who Live With a Cat
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R1908-1909-ALG-2102; 2021-002089-42 (EudraCT Number)
Record Dates: First submitted 2021-07-19; First posted 2021-07-29 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-05

CONDITIONS: Allergic Rhinitis Due to Cat Allergy
Keywords: Cat allergy induced allergic rhinitis; Allergic conjunctivitis; Asthma
MeSH Terms: conditions — Conjunctivitis, Allergic; Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- REGN1908-1909 (Experimental): Randomized 1:1
  Interventions: Drug: REGN1908-1909
- Placebo (Placebo Comparator): Randomized 1:1
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: REGN1908-1909 — Subcutaneous (SC) for a total of 5 administrations
  Arms: REGN1908-1909
Drug: Matching Placebo — SC for a total of 5 administrations
  Arms: Placebo

SUMMARY:
The primary objective of the study is to determine the efficacy of REGN1908-1909, as compared to placebo, to reduce allergic rhinitis/conjunctivitis symptoms and allergy rescue medication use during natural cat exposure.

The Secondary Objectives are:

* To assess the reduction of allergic symptoms and use of allergy rescue medications after treatment with REGN1908-1909 versus placebo, as measured by the individual components of the CSMS
* To assess health-related quality of life (HRQoL) as measured by the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ[S])
* To determine the efficacy of REGN1908-1909, as compared to placebo, to inhibit a wheal-and-flare response to a skin prick test with cat allergen
* To assess the durability of effect in allergic rhinitis and conjunctivitis symptom and medication scores after multiple doses of REGN1908-1909 compared to placebo given every 12 weeks (Q12W)
* To determine the efficacy following multiple doses of REGN1908-1909 compared to placebo at inhibiting a wheal-and-flare response to a skin prick test with cat allergen
* To estimate the effect of REGN1908-1909 on lung function, as compared to placebo, in patients with asthma
* To determine the efficacy of REGN1908-1909 as compared to placebo to reduce asthma symptoms in patients with asthma
* To assess whether there is a difference in asthma rescue medication use in patients with asthma who are treated with REGN1908-1909 compared to placebo
* To assess whether there is a difference in nighttime awakenings in patients with asthma treated with REGN1908-1909 compared to placebo
* To evaluate the short-term and long-term safety and tolerability of REGN1908-1909, including the incidence of hypersensitivity reactions, local injection site reactions, and asthma exacerbations
* To determine systemic exposure of total (free and antigen-bound) antibodies as measured by concentration of REGN1908 and REGN1909
* To assess the immunogenicity of REGN1908 and REGN1909

ELIGIBILITY:
Key Inclusion Criteria:

1. Generally healthy males and females who are 12 years and older at the time of screening.
2. Weight must be ≥40 kg at the time of screening
3. Documented or patient reported history (for at least 2 years) of symptomatic cat allergen-triggered allergic rhinitis with or without conjunctivitis and with or without asthma as defined by all of the following criteria:

   1. Positive skin prick test (SPT) with cat hair extract (mean wheal diameter at least 5 mm greater than a negative control) at screening
   2. Positive allergen-specific IgE (sIgE) tests for cat and Fel d 1 (both ≥0.7 kUa/L at screening)
   3. Documented or patient reported history of nasal and/or ocular symptoms upon cat exposure
   4. Symptomatic despite the use of medications to treat their nasal and/or ocular symptoms
4. At least 1 generally healthy cat (that is unlikely to die during the study) living in the home resulting in regular exposure
5. A daily total rhinitis/conjunctivitis symptom score (total symptom score [TSS]) of at least 8 of 18 during at least 8 days of the 15-day baseline assessment period and use of standard, therapeutic doses of pharmacotherapy for the treatment of allergic rhinoconjunctivitis on at least 8 days of the 15-day baseline assessment period.

Key Exclusion Criteria:

1. History of significant multiple and/or severe allergies, as assessed by the investigator, that would potentially interfere with the assessments during the baseline and 12-week efficacy assessment periods or confound results, per investigator discretion, including significant rhinitis or sinusitis due to daily contact with other allergens causing symptoms that are expected to coincide with the baseline period or any of the efficacy assessment periods
2. Received REGN1908-1909 in a prior REGN1908-1909 clinical trial (receipt of placebo in a previous trial is allowed)
3. Active lung disease other than asthma
4. FEV1 less than 70% of predicted at screening or randomization
5. Treatment with an investigational drug within 2 months or within 5 half-lives (if known), whichever is longer, prior to screening
6. Persistent chronic or recurring acute infection requiring treatment with antibiotics, antivirals, or antifungals, or any untreated respiratory infections within 4 weeks prior to screening. Patients may be re-evaluated after resolution of symptoms and specified time duration

NOTE: Other protocol-defined Inclusion/ Exclusion Criteria apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (92):
- United States (42):
  - Allergy and Asthma Associates of Southern California - CRN - PPDS, Mission Viejo, California
  - Integrated Research of Inland, Inc, Riverside, California
  - Peninsula Research Associates - CRN - PPDS, Rolling Hills Estates, California
  - Allergy and Asthma Medical Group and Research Center - CRN - PPDS, San Diego, California
  - Asthma and Allergy Associates PC - CRN - PPDS, Colorado Springs, Colorado
  - Colorado Allergy and Asthma Centers PC - CRN - PPDS, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - Velocity Clinical Research, Inc. (Meridan), Meridian, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Asthma and Allergy Center of Chicago Sc-Oak Park, Oak Park, Illinois
  - Sneeze Wheeze and Itch Associates LLC, Springfield, Illinois
  - South Bend Clinic, South Bend, Indiana
  - Bluegrass Allergy Research, Lexington, Kentucky
  - Allergy and Asthma Specialists PSC, Owensboro, Kentucky
  - Charleston Allergy and Asthma, Baltimore, Maryland
  - Institute For Asthma and Allergy, Chevy Chase, Maryland
  - Respiratory Medicine Research Institute of Michigan PLC, Ypsilanti, Michigan
  - Clinical Research Institute, Inc - CRN - PPDS, Plymouth, Minnesota
  - University of Missouri - Hospital, Columbia, Missouri
  - Montana Medical Research, Missoula, Montana
  - Somnos Clinical Research, Lincoln, Nebraska
  - Nebraska Medical Research Institute, Inc. - CRN - PPDS, Papillion, Nebraska
  - Riverside Medical Group - Circuit - PPDS, Belleville, New Jersey
  - Atlantic Research Center LLC, Ocean City, New Jersey
  - Princeton Center For Clinical Research - CRN - PPDS, Skillman, New Jersey
  - Allergy Partners of NJ, P.C., Teaneck, New Jersey
  - Allergy Consultants PA, Verona, New Jersey
  - SUNY Downstate Health Science University, Brooklyn, New York
  - NYU Langone Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Allergy Partners of Western North Carolina, Asheville, North Carolina
  - Bernstein Clinical Research Center Inc, Cincinnati, Ohio
  - Optimed Research Ltd - Clinedge - PPDS, Columbus, Ohio
  - Aventiv Research Inc - Columbus - HyperCore - PPDS, Dublin, Ohio
  - Allergy Asthma and Clinical Research Center, Oklahoma City, Oklahoma
  - PDX Allergy, LLC dba Portland Research, Happy Valley, Oregon
  - Northwest Research Center - CRN - PPDS, Portland, Oregon
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - Asthma, Nasal Disease and Allergy Research Center of New England, East Providence, Rhode Island
  - Asthma & Allergy Physicians of Rhode Island Clinical Research Institute (AAPRI CRI), Warwick, Rhode Island
  - Seattle Allergy & Asthma Research Institute, Seattle, Washington
  - The Medical College of Wisconsin, Inc., Greenfield, Wisconsin
- Belgium (4):
  - UZ Gent, Ghent, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams Brabant
  - Private Practice Dr Jean Benoit Martinot, Erpent
  - CHR de la Citadelle, Liège
- Canada (11):
  - Aggarwal and Associates Ltd, Brampton, Ontario
  - Hamilton Allergy, Hamilton, Ontario
  - Kingston Health Science Centre, Kingston, Ontario
  - Red Maple Trials, Ottawa, Ontario
  - Stouffville Medical Clinic, Stouffville, Ontario
  - Gordon Sussman Clinical Research Inc, Toronto, Ontario
  - Toronto Allergy Clinic, Toronto, Ontario
  - Joel Liem Medicine Professional Corporation, Windsor, Ontario
  - LMC Manna Research - Quebec - HyperCore - PPDS, Lévis, Quebec
  - Centre d'investigation Clinique Mauricie, Trois-Rivières, Quebec
  - Clinique Spécialisée en Allergie de la Capitale, Québec
- Nouvel Hopital Civil, Strasbourg, Bas-Rhin, France
- Germany (14):
  - HNO Praxis am Neckar, Heidelberg, Baden-Wurttemberg
  - Klinikum Stuttgart, Stuttgart, Baden-Wurttemberg
  - Beldio Research GmbH, Memmingen, Bavaria
  - Praxis Dr. med. Elke Decot, Dreieich, Hesse
  - Praxis Dr. med. Claus Keller, Frankfurt am Main, Hesse
  - Praxis Dr. med. Gerhard Schindlbeck, Viernheim, Hesse
  - Universitatsklinikum Munster, Münster, North Rhine-Westphalia
  - Klinische Forschung Dresden GmbH (KFGN), Dresden, Saxony
  - Praxis für HNO und Allergologie, Dresden, Saxony
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden, Saxony
  - Salvus-Klinische Studien GmbH, Leipzig, Saxony
  - BAG Prof. Dr. G. Hoheisel Dr. A. Bonitz, Leipzig, Saxony
  - Charité - Universitätsmedizin Berlin, Berlin
  - Emovis GmbH, Berlin
- Poland (20):
  - Centrum Alergologii Teresa Hofman, Piła, Greater Poland Voivodeship
  - Centrum Nowoczesnych Terapii Dobry Lekarz Sp. z o.o., Krakow, Lesser Poland Voivodeship
  - Alergo-Med Specjalistyczna Przychodnia Lekarska Sp. z.o.o, Tarnów, Lesser Poland Voivodeship
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - ALL-MED - Specjalistyczna Opieka Medyczna - Medyczny Instytut Badawczy, Wroclaw, Lower Silesian Voivodeship
  - ETG Lublin - PPDS, Lublin, Lublin Voivodeship
  - Centrum Alergologii Specjalistyczna Przychodnia Alergologiczna, Lublin, Lublin Voivodeship
  - ETG Zamosc - PPDS, Zamość, Lublin Voivodeship
  - Malopolskie Centrum Alergologii, Krakow, Malopolski
  - ETG Warszawa - PPDS, Piaseczno, Masovian Voivodeship
  - EMed Centrum Uslug Medycznych, Rzeszów, Podkarpackie Voivodeship
  - Homeo Medicus Szczesiul sp. j., Bialystok, Podlaskie Voivodeship
  - Clinica Vitae Sp z o o, Gdansk, Pomeranian Voivodeship
  - Specjalistyczna Przychodnia Lekarska Alergo-Med Sp. z.o.o, Poznan
  - SPZOZ Uniwersytecki Szpital Kliniczny nr 1 im Norberta Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz, Łódź Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Wojskowej Akademii Medycznej Centralny Szpital Weteranow, Lodz, Łódź Voivodeship
  - ETG Lodz - PPDS, Lodz, Łódź Voivodeship
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Lodz, Łódź Voivodeship
  - IP Clinic Sp. z o. o., Lodz, Łódź Voivodeship
  - ETG Kielce, Kielce, Świętokrzyskie Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1,227 participants were screened, 446 participants were randomized
Groups:
- Placebo: Randomized 1:1 ratio of matching placebo for REGN1908-1909 600 mg administered Q12W for a total of 5 administrations
- REGN1908-1909: Randomized 1:1 ratio of REGN1908-1909 600 mg administered Q12W for a total of 5 administrations
Period: Overall Study
Arm/Group | Placebo | REGN1908-1909
Started | 222 | 224
Completed | 8 | 4
Not Completed | 214 | 220
Not completed — Protocol Violation | 0 | 3
Not completed — Adverse Event | 1 | 3
Not completed — Pregnancy | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Sponsor Request | 157 | 172
Not completed — Lost to Follow-up | 4 | 5
Not completed — Withdrawal by Subject | 50 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | REGN1908-1909 | Total
Number analyzed (Participants) | 222 | 224 | 446
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (12.68) | 37.4 (12.58) | 37.2 (12.62)
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0
  Children (2-11 years) | 0 | 0 | 0
  Adolescents (12-17 years) | 8 | 6 | 14
  Adults (18-64 years) | 211 | 215 | 426
  From 65-84 years | 3 | 3 | 6
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 147 | 283
  Male | 86 | 77 | 163
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 7 | 11 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 210 | 206 | 416
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 2 | 1 | 3
Ethnicity [Count of Participants; unit: Participants]
  NOT HISPANIC OR LATINO | 216 | 217 | 433
  HISPANIC OR LATINO | 5 | 5 | 10
  NOT REPORTED | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Daily Combined Symptom and Medication Score (CSMS) Averaged Over Last 12 Weeks of the Treatment Period in Patients Who Receive REGN1908-1909 Versus Placebo
Description: CSMS is calculated by adding the Daily Medication Score (DMS) and Total Symptom Score (TSS) together, with scores ranging between 0 (none) and 38 (severe).
Time Frame: Weeks 48 to 60
Population: Due to the early termination, the study was not fully enrolled, the primary endpoint and all secondary endpoints planned for weeks 48 - 60 could not be evaluated. Data not collected.
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Daily Total Nasal Symptom Score (TNSS) Averaged Over the Last 12 Weeks of Treatment Period in Patients Who Receive REGN1908-1909 Versus Placebo
Description: Total nasal symptom score (TNSS) is from 0 to 12 and is based on assessment of 4 nasal symptoms graded on a Likert scale ranging from 0 (none) to 3 (severe) for congestion, itching, and rhinorrhea, and from 0 (none) to 3 (5 or more sneezes) for sneezing.
Time Frame: Weeks 48 to 60
Population: as for outcome 1
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percent Change From Pre-treatment Baseline in Average CSMS Over the Last 12 Weeks of the Treatment Period in Patients Who Receive REGN1908-1909 Versus Placebo
Time Frame: Weeks 48 to 60
Population: as for outcome 1
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percent Change From Pre-treatment Baseline in Average TNSS Over the Last 12 Weeks of the Treatment Period in Patients Who Receive REGN1908-1909 Versus Placebo
Time Frame: Weeks 48 to 60
Population: as for outcome 1
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Daily Total Symptom Score (TSS) Averaged Over the Last 12 Weeks of the Treatment Period in Patients Who Receive REGN1908-1909 Versus Placebo
Description: TSS is a combined score of TOSS and TNSS. TNSS and TOSS are scored as in part 1 each for a combined TSS of 0 (none) to 18 (severe)
Time Frame: Weeks 48 to 60
Population: as for outcome 1
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percent Change From Pre-treatment Baseline in Average TSS Over the Last 12 Weeks of the Treatment Period in Patients Who Receive REGN1908-1909 Versus Placebo
Time Frame: Weeks 48 to 60
Population: as for outcome 1
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percent Change From Baseline to the End of Treatment in Cat Skin Prick Test (SPT) Mean Wheal Diameter in Patients Who Receive REGN1908-1909 Versus Placebo
Time Frame: Week 60
Population: as for outcome 1
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Daily CSMS Averaged Over the Initial 12 Weeks of the Treatment Period in Patients Who Receive REGN1908-1909 Versus Placebo
Description: The combined symptom and medication score (CSMS) is defined as the daily combined allergic rhinitis and conjunctivitis total symptom score (TSS: calculated as the sum of total nasal symptom score [TNSS] and total ocular symptom score [TOSS]) plus daily medication score (DMS). Scores ranging between 0 (none) and 38 (severe).
Time Frame: Weeks 0 to 12
Population: The full analysis set (FAS) includes all randomized patients; it is based on the treatment allocated (as randomized). Efficacy endpoints will be analyzed using the FAS.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 224 | 222
Scores on a Scale | 16.184 (0.9370) [lower limit 0.9370] | 15.290 (0.9173) [lower limit 0.9173]

9. Secondary Outcome: Daily TNSS Averaged Over the Initial 12 Weeks of the Treatment Period in Patients Who Receive REGN1908-1909 Versus Placebo
Description: The TNSS ranges from 0 to 12 and is based on assessment of 4 nasal symptoms graded on a Likert scale ranging from 0 (none) to 3 (severe) for nasal congestion, itching, and runny nose, and sneezing.
Time Frame: Weeks 0 to 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Average Score
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 224 | 222
Average Score | 6.18 (0.320) [lower limit 0.320] | 5.88 (0.314) [lower limit 0.314]

10. Secondary Outcome: Percent Change From Pre-treatment Baseline in Average CSMS Over the Initial 12 Weeks of the Treatment Period in Patients Who Receive REGN1908-1909 Versus Placebo
Description: The combined symptom and medication score (CSMS) is defined as the daily combined allergic rhinitis and conjunctivitis total symptom score (TSS: calculated as the sum of total nasal symptom score [TNSS] and total ocular symptom score [TOSS]) plus daily medication score (DMS).
Time Frame: Weeks 0 to 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 224 | 222
Percent Change | -29.25 (4.363) [lower limit 4.363] | -33.16 (28.299) [lower limit 28.299]

11. Secondary Outcome: Percent Change From Pre-treatment Baseline in Average TNSS Over the Initial 12 Weeks of the Treatment Period in Patients Who Receive REGN1908-1909 Versus Placebo
Description: as for outcome 9
Time Frame: Weeks 0 to 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 224 | 222
Percent Change | -26.77 (29.471) [lower limit 29.471] | -30.33 (27.976) [lower limit 27.976]

12. Secondary Outcome: Percent Change From Pre-treatment Baseline in Average TSS Over the Initial 12 Weeks of the Treatment Period in Patients Who Receive REGN1908-1909 Versus Placebo
Description: Total symptom score (TSS: calculated as the sum of TNSS and total ocular symptom score [TOSS]) plus daily medication score (DMS).
Time Frame: Weeks 0 to 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 224 | 222
Percent | -27.25 (30.185) [lower limit 30.185] | -31.16 (28.390) [lower limit 28.390]

13. Secondary Outcome: Daily TSS Score Averaged Over the Initial 12 Weeks of the Treatment Period in Patients Who Receive REGN1908-1909 Versus Placebo
Description: as for outcome 12
Time Frame: Weeks 0 to 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Average Score
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 224 | 222
Average Score | 8.11 (3.743) [lower limit 3.743] | 7.80 (3.507) [lower limit 3.507]

14. Secondary Outcome: Percent Change From Pre-treatment Baseline in Average TOSS, Over the Initial 12 Weeks of the Treatment Period in Patients Who Receive REGN1908-1909 Versus Placebo
Description: Total ocular symptom score is 0 to 6 and is based on itching/redness/gritty feeling and tearing/watering; each of the 2 symptoms is graded 0 (absent), 1 (mild), 2 (moderate), and 3 (severe)
Time Frame: Weeks 0 to 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 224 | 222
Percent Change | -27.90 (38.216) [lower limit 38.216] | -32.92 (35.708) [lower limit 35.708]

15. Secondary Outcome: Daily TOSS Averaged Over the Last 12 Weeks of the Treatment Period in Patients Who Receive REGN1908-1909 Versus Placebo
Description: as for outcome 14
Time Frame: Weeks 48 to 60
Population: as for outcome 1
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Percent Change From Pre-treatment Baseline in Average TOSS Over the Last 12 Weeks of the Treatment Period in Patients Who Receive REGN1908-1909 Versus Placebo
Description: as for outcome 14
Time Frame: Weeks 48 to 60
Population: as for outcome 1
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Percent Change in Forced Expiratory Volume (FEV)1 in Patients With Asthma Who Receive REGN1908-1909 Versus Placebo
Description: In-clinic spirometry on all patients to determine FEV1 (forced expiratory volume in 1 second) in liters (L).
Time Frame: Baseline to week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 117 | 112
Percent Change | 1.35 (7.314) [lower limit 7.314] | -0.05 (5.334) [lower limit 5.334]

18. Secondary Outcome: Percent Change in FEV1 in Patients With Asthma Who Receive REGN1908-1909 Versus Placebo
Description: In-clinic spirometry on all patients to determine FEV1 (forced expiratory volume in 1 second) in liters (L).
Time Frame: Baseline to week 60
Population: as for outcome 1
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Percent Change in Cat SPT Mean Wheal Diameter in Patients Who Receive REGN1908-1909 Versus Placebo
Description: The full analysis set (FAS) includes all randomized participants; it is based on the treatment allocated (as randomized). Efficacy endpoints will be analyzed using the FAS.
Time Frame: Baseline to week 72
Population: as for outcome 1
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Daily Number of Nighttime Awakenings Averaged Over the Initial 12 Weeks of the Treatment Period in Patients With Asthma Who Receive REGN1908-1909 Versus Placebo
Time Frame: Weeks 0 to 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Nighttime awakenings/Day
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 117 | 112
Nighttime awakenings/Day | 0.54 (0.846) [lower limit 0.846] | 0.72 (1.166) [lower limit 1.166]

21. Secondary Outcome: Number of Participants With Adverse Event of Special Interests (AESIs) Throughout the Study
Time Frame: Weeks 0 to 72
Measure: Number; unit: Participants
Arm/Group | Placebo | REGN1908-1909
Number analyzed (Participants) | 222 | 224
Participants | 0 | 2

22. Secondary Outcome: Number of Participants With Serious Treatment-Emergent Adverse Events (TEAEs) Throughout the Study
Time Frame: Weeks 0 to 60
Measure: Number; unit: Participants
Arm/Group | Placebo | REGN1908-1909
Number analyzed (Participants) | 222 | 224
Participants | 2 | 2

23. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Throughout the Study
Time Frame: Weeks 0 to 72
Measure: Number; unit: Participants
Arm/Group | Placebo | REGN1908-1909
Number analyzed (Participants) | 222 | 224
Participants | 2 | 2

24. Secondary Outcome: Total REGN1908 Concentration in Serum Over the Study Duration
Time Frame: Weeks 0 to 60
Population: Each PK analysis includes all treated participants who received any amount of study drug (active, [SAF]) and had at least 1 non-missing result of each respective analyte following the first dose of study drug. The PKAS is based on the actual treatment received (as treated) rather than as randomized. Placebo participants were not analyzed.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | REGN1908-1909
Number analyzed (Participants) | 224
mg/L
  Baseline [12 years old < 18 years old]: number analyzed (Participants) | 6
  Baseline [12 years old < 18 years old] | 0.0753 (0.123)
  Week 12 [12 years old < 18 years old]: number analyzed (Participants) | 5
  Week 12 [12 years old < 18 years old] | 7.19 (2.54)
  Week 24 [12 years old < 18 years old]: number analyzed (Participants) | 4
  Week 24 [12 years old < 18 years old] | 10.5 (2.04)
  Week 36 [12 years old < 18 years old]: number analyzed (Participants) | 4
  Week 36 [12 years old < 18 years old] | 9.56 (4.98)
  Baseline ( >= 18 years old): number analyzed (Participants) | 205
  Baseline ( >= 18 years old) | 0.0179 (0.116)
  Week 12 ( >= 18 years old) 3: number analyzed (Participants) | 193
  Week 12 ( >= 18 years old) 3 | 5.26 (2.60)
  Week 24 ( >= 18 years old): number analyzed (Participants) | 169
  Week 24 ( >= 18 years old) | 5.99 (3.58)
  Week 36 ( >= 18 years old): number analyzed (Participants) | 126
  Week 36 ( >= 18 years old) | 4.47 (3.63)
  Week 48 ( >= 18 years old): number analyzed (Participants) | 67
  Week 48 ( >= 18 years old) | 2.14 (2.76)
  Week 60 ( >= 18 years old): number analyzed (Participants) | 11
  Week 60 ( >= 18 years old) | 0.526 (0.377)

25. Secondary Outcome: Total REGN1909 Concentration in Serum Over the Study Duration
Time Frame: Weeks 0 to 60
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | REGN1908-1909
Number analyzed (Participants) | 224
mg/L
  Baseline [12 years old < 18 years old]: number analyzed (Participants) | 6
  Baseline [12 years old < 18 years old] | 0 (0)
  Week 12 [12 years old < 18 years old]: number analyzed (Participants) | 5
  Week 12 [12 years old < 18 years old] | 3.49 (1.99)
  Week 24 [12 years old < 18 years old]: number analyzed (Participants) | 4
  Week 24 [12 years old < 18 years old] | 4.59 (0.957)
  Week 36 [12 years old < 18 years old]: number analyzed (Participants) | 4
  Week 36 [12 years old < 18 years old] | 4.02 (2.39)
  Baseline [>= 18 years old]: number analyzed (Participants) | 205
  Baseline [>= 18 years old] | 0.0160 (0.118)
  Week 12 [>= 18 years old]: number analyzed (Participants) | 193
  Week 12 [>= 18 years old] | 2.32 (1.50)
  Week 24 [>= 18 years old]: number analyzed (Participants) | 169
  Week 24 [>= 18 years old] | 2.46 (1.79)
  Week 36 [>= 18 years old]: number analyzed (Participants) | 126
  Week 36 [>= 18 years old] | 1.91 (2.03)
  Week 48 [>= 18 years old]: number analyzed (Participants) | 67
  Week 48 [>= 18 years old] | 0.903 (1.47)
  Week 60 [>= 18 years old]: number analyzed (Participants) | 11
  Week 60 [>= 18 years old] | 0.161 (0.175)

26. Secondary Outcome: Incidence of Treatment-emergent Anti-drug Antibodies (ADAs) to REGN1908 Throughout the Study
Time Frame: Weeks 0 to 72
Population: The AAS is defined for each study drug separately and includes all treated participants who received any amount of study drug (active or placebo, [SAF]) and had at least 1 non-missing ADA result following the first dose of study drug or placebo. The AAS is based on the actual treatment received (as treated) rather than as randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 210 | 213
Participants | 6 | 4

27. Secondary Outcome: Incidence of Treatment-emergent ADAs to REGN1909 Throughout the Study
Time Frame: Weeks 0 to 72
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 210 | 213
Participants | 5 | 5

28. Secondary Outcome: Percent Change in Cat SPT Mean Wheal Diameter in Patients Who Receive REGN1908-1909 Versus Placebo (up to Week 12)
Time Frame: Baseline to week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 224 | 222
Percent Change | -35.27 (31.438) [lower limit 31.438] | -26.76 (33.787) [lower limit 33.787]

29. Secondary Outcome: Percent Change in FEV1 in Participants With Asthma Who Receive REGN1908-1909 Versus Placebo (up to Week 12)
Time Frame: Baseline to week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 224 | 222
Percent Change | 0.0321 (0.21546) [lower limit 0.21546] | -0.0086 (0.17005) [lower limit 0.17005]

30. Secondary Outcome: Percent Change in FEV1 in Participants With Asthma Who Receive REGN1908-1909 Versus Placebo (up to Week 60)
Time Frame: Baseline to week 60
Population: as for outcome 1
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Change From Baseline to Week 60 in Rhinoconjunctivitis Quality of Life Questionnaire for Ages 12+ (RQLQ(S)+12) in Participants Who Received REGN1908-1909 Versus Placebo
Description: The RQLQ had 25 questions in 6 domains (nose symptoms, eye symptoms, practical problems, activity limitation, non-hay fever symptoms and emotional function). Participants recalled how they have been during the previous week and responded to each question on a 7-point scale. The overall RQLQ score was the mean of all 25 responses and the individual domain scores were the means of the items in those domains. The RQLQ(S) responses are based on a 7-point Likert scale with responses ranging from 0 (not troubled) to 6 (extremely troubled).
Time Frame: Baseline to week 60
Population: as for outcome 1
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Daily Medication Score (DMS) Averaged Over the Initial 12 Weeks of the Treatment Period in Participants Who Receive REGN1908-1909 Versus Placebo
Description: The Daily Medication Score (DMS) was calculated by adding points for each pre-specified medication. Participants will be asked to record their daily rescue medication use using an e-diary, including which medications and the amount of these prespecified medications. The scale is 0 (minimum) to 20 (maximum)
Time Frame: Weeks 0 to 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 224 | 222
Score on a scale | 6.582 (4.9101) [lower limit 4.9101] | 6.467 (4.5117) [lower limit 4.5117]

33. Secondary Outcome: DMS Averaged Over the Last 12 Weeks of the Treatment Period in Participants Who Receive REGN1908-1909 Versus Placebo
Time Frame: Weeks 48 to 60
Population: as for outcome 1
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: Percent Change From Pre-treatment Baseline in Average DMS Averaged Over the Last 12 Weeks of the Treatment Period in Participants Who Receive REGN1908-1909 Versus Placebo
Time Frame: Weeks 48 to 60
Population: as for outcome 1
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Asthma Daily Symptom (ADS) Score, Averaged Over the Initial 12 Weeks of the Treatment Period Using Asthma Daytime Symptom Diary (ADSD) and the Asthma Nighttime Symptom Diary (ANSD) in Participants With Asthma Who Receive REGN1908-1909 Versus Placebo
Description: The total daily asthma symptom score is a participant-reported outcome concerning the occurrence of asthma symptoms and their effect on a patient's daily activities and sleep. It is composed of two parts: daytime (five items) and nighttime (four items), both scored ordinally. Higher scores indicate more severe symptoms. The ADSD score will be based on 6 patient-reported symptoms (difficulty breathing, wheezing, shortness of breath, chest tightness, chest pain, and cough at their worst using an 11-point numeric rating scale (NRS) ranging from 0 ('None') to 10 ('As bad as you can imagine').
Time Frame: Weeks 0 to 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 117 | 112
Score on a scale | 2.17 (2.005) [lower limit 2.005] | 2.52 (2.141) [lower limit 2.141]

36. Secondary Outcome: ADS Score Averaged Over the Last 12 Weeks of the Treatment Period Using ADSD and the ANSD in Participants With Asthma Who Receive REGN1908-1909 Versus Placebo (Weeks 48 to 60)
Time Frame: Weeks 48 to 60
Population: as for outcome 1
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 0 | 0

37. Secondary Outcome: Daily TOSS Averaged Over the Initial 12 Weeks of the Treatment Period in Participants Who Receive REGN1908-1909 Versus Placebo
Description: The TOSS ranges from 0 to 6 and is based on 2 eye symptoms: itching/redness/gritty feeling and tearing/watering. Each of the 2 symptoms is graded on a Likert scale ranging from 0 (none) to 3 (severe).
Time Frame: Weeks 0 to 12
Population: The full analysis set (FAS) includes all randomized patrticipants; it is based on the treatment allocated (as randomized). Efficacy endpoints will be analyzed using the FAS.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 224 | 222
Score on a scale | 2.42 (1.414) [lower limit 1.414] | 2.33 (1.346) [lower limit 1.346]

38. Secondary Outcome: Change From Baseline to Week 60 in Asthma Control Questionnaire 5 Question Version (ACQ-5) in Participant With Asthma Who Receive REGN1908-1909 Versus Placebo
Description: The ACQ-5 had 5 questions, reflecting the top-scoring five asthma symptoms: woken at night by symptoms, wake in the mornings with symptoms, limitation of daily activities, shortness of breath and wheeze. Participants were asked to recall how their asthma had been during the previous week and to respond to each of the five symptom questions on a 7-point scale ranged from 0 (no impairment) to 6 (maximum impairment). ACQ-5 total mean score was mean of the scores of all 5 questions and, therefore, ranged from 0 (totally controlled) to 6 (severely uncontrolled), higher scores indicated lower asthma control.
Time Frame: Baseline to week 60
Population: as for outcome 1
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 0 | 0

39. Secondary Outcome: Daily Number of Nighttime Awakenings Averaged Over the Last 12 Weeks of the Treatment Period in Patients With Asthma Who Receive REGN1908-1909 Versus Placebo (Weeks 48 to 60)
Time Frame: Weeks 48 to 60
Population: as for outcome 1
Arm/Group | REGN1908-1909 | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose to study termination (~60 weeks)
Groups:
- R1908-1909 600 mg: Randomized 1:1 ratio of REGN1908-1909 600 mg administered Q12W for a total of 5 administrations
Arm/Group | Placebo | R1908-1909 600 mg
All-Cause Mortality (participants affected / at risk) | 0/222 | 0/218
Serious Adverse Events (participants affected / at risk) | 2/222 | 2/218
Other Adverse Events (participants affected / at risk) | 58/222 | 54/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=222) | R1908-1909 600 mg (N=218)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=222) | R1908-1909 600 mg (N=218)
COVID-19 (Infections and infestations) | 28 (29) | 22 (22)
Nasopharyngitis (Infections and infestations) | 25 (30) | 21 (28)
Upper respiratory tract infection (Infections and infestations) | 9 (11) | 14 (16)

LIMITATIONS AND CAVEATS:
The study met prespecified interim futility criteria for CSMS and TNSS, therefore, an efficacy analysis was not performed for the primary and secondary endpoints as specified in the protocol

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT04981717/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT04981717/SAP_001.pdf